CLINICAL TRIAL: NCT02651298
Title: Fractional CO2-laser Treatment of Caesarean Section Scars - A Randomized Controlled Split-scar Trial With Long Term Follow-up Assessment
Brief Title: CO2-laser Treatment for Caesarean Section Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Lumenis Be Ltd. (Industry)
Responsible Party: Principal Investigator, Katrine Elisabeth Karmisholt, MD, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-section
Record Dates: First submitted 2016-01-02; First posted 2016-01-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Cicatrix
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fractional CO2-laser (Experimental): 3 treatments with fractional co2-laser
  Interventions: Device: Fractional Co2-laser
- Untreated control (No Intervention): untreated control side of caesarean section scar

INTERVENTIONS:
Device: Fractional Co2-laser — laser treatment
  Other Names: Ablative fractional laser
  Arms: Fractional CO2-laser

SUMMARY:
Fractional Co2-laser for treatment of mature caesarean section scars.

DETAILED DESCRIPTION:
Randomized split scar study to document improvement of caesarean section scars as compared to untreated control scar.

ELIGIBILITY:
Inclusion Criteria:

* mature caesarean section scar

Exclusion Criteria:

* systemic uncontrolled disease
* recent or current cancer
* smoking
* keloid formation
* wounds or local disease int treatment area
* pregnancy or lactation

Ages: 22 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
patient observer scar scale | up until 6 months post treatment
  validated scar scale evaluations

SECONDARY OUTCOMES:
erythema measured by reflectance | 1 months post treatment
  measured by reflectance
pigmentation measured by reflectance | 1 months post treatment
  measured by reflectance
erythema measured by reflectance | 3 months post treatment
  measured by reflectance
pigmentation measured by reflectance | 3 months post treatment
  measured by reflectance
erythema measured by reflectance | 6 months post treatment
  measured by reflectance
pigmentation measured by reflectance | 6 months post treatment
  measured by reflectance
histology of scar tissue | 3 months post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Merete Haedersdal, Professor, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark